CLINICAL TRIAL: NCT04120922
Title: The Effect of Calcium-based and Calcium-free Phosphate-binders on Bone Mineral Content, Measured by a Novel Technique of Dual-tracer Stable Calcium Isotope Method, in Children With Chronic Kidney Disease or on Dialysis - a Time Series Trial
Brief Title: Assessing Bone Calcium Content in Children With Kidney Disease Treated With Two Different Medicines
Acronym: CAL-BAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTU/2014/146; CDF-2016-09-038 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2019-09-18; First posted 2019-10-09 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Diseases
Keywords: Dialysis; chronic kidney disease stage 3b, 4-5; calcium isotope ratio; bone mineral content; Calcium isotope fractions δ44/42Ca
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Calcium Carbonate; Sevelamer

STUDY DESIGN:
Intervention Model Description: A open label, time series trial
Masking Description: This is a time series open label trial so there is no randomisation or blinding to treatment. All analyses will be performed in a blinded manner and the treating clinicians will be blinded to the results of the calcium isotope ratios until after participants have completed their trial related administration of P-binder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium carbonate (Other): Calcium based P-binder - calcium carbonate: Typical dose is 500mg, orally, three times a day but this can be adjusted as per individual patient requirements at the clinician's discretion.
  All participants will be given sevelamer carbonate (Ca-free P-binder) for up to 16 weeks and then calcium carbonate (Ca-based P-binder) for 12 weeks, administered orally. No wash out period is possible as the children must always be on a P-binder. The Ca-free P-binder may be administered for less than 16 weeks if it is clinically necessary to resume the Ca-based P-binder early based on serial monitoring of serum Ca levels.
  Interventions: Other: calcium carbonate; Other: sevelamer carbonate
- sevelamer carbonate (Other): Calcium (Ca) free P-binder - sevelamer carbonate: Typical dose is 800mg, orally, three times a day but this can be adjusted as per individual patient requirements at the clinician's discretion.
  All participants will be given sevelamer carbonate (Ca-free P-binder) for up to 16 weeks and then calcium carbonate (Ca-based P-binder) for 12 weeks, administered orally. No wash out period is possible as the children must always be on a P-binder. The Ca-free P-binder may be administered for less than 16 weeks if it is clinically necessary to resume the Ca-based P-binder early based on serial monitoring of serum Ca levels.
  Interventions: Other: calcium carbonate; Other: sevelamer carbonate

INTERVENTIONS:
Other: calcium carbonate — See arm description
Other: sevelamer carbonate — See arm description

SUMMARY:
This is an open label, time series trial. The trial is likely to be single centre (additional sites will only be opened if necessary) and will involve 25 children with chronic kidney disease (stage 3b, 4-5) or on dialysis. The overall aim of this trial is to explore the viability of the Ca isotope ratio measured by dual-tracer stable Ca isotope method as a measure of bone mineral (Ca) content, and to evaluate how it changes in response to two commonly used medications that either contain Ca (calcium carbonate) or do not (sevelamer carbonate). Both calcium carbonate and sevelamer carbonate are routinely used in children, but their effect on the bone mineral content (measured by the Ca isotope ratio) has not been studied.

This short-term trial will provide proof-of-concept data to determine the utility of the Ca isotope fractionation technique in guiding medication usage in children with CKD and on dialysis. These data will inform a potential future randomised trial that utilises the calcium isotope fractionation technique to adjust the calcium intake (through diet and different medications, including vitamin D analogues) and monitor changes in important patient level outcomes such as fractures and bone mineral density on DXA scan.

Participants will be administered sevelamer carbonate first for 16 weeks and then will switch to calcium carbonate for 12 weeks. Participants may need to change medication earlier than 16 weeks at the clinician's discretion based on their calcium levels on routine blood tests.

Calcium isotope levels will be measured in blood and urine samples for up to 28 weeks. Isotopes levels in faeces and dialysis fluid samples may also be measured.

This is not a Clinical Trial of an Investigational Medicinal Product (CTIMP).

DETAILED DESCRIPTION:
Lay Summary of Background and Rationale:

The growing bones of children need calcium in order to mineralise (become strong). Children with kidney failure (called chronic kidney disease; CKD) or on dialysis can often be calcium deficient. They are given medications with extra calcium to help their bones mineralise. However, there is currently no practical way of measuring bone mineralisation. Doctors may perform special x-rays, but it takes many months before any bone structure problems become apparent on X-rays. Doctors giving children additional calcium do not know how much to give. Sometimes children are given too little and their bones do not mineralise adequately, or they are given too much, and the excess calcium is deposited in their arteries causing vascular calcification. Timely and practical ways of measuring bone mineralisation are needed so doctors can accurately determine the amount of calcium containing medicines they give.

The CAL-BAL trial will evaluate a novel potential biomarker of bone mineralisation: the calcium isotope ratio (δ44/42Ca) which will be measured in blood and urine. The trial will collect information on δ44/42Ca for patients with CKD or on dialysis for 28 weeks. It will measure how δ44/42Ca changes when a patient switches from a medicine containing calcium to one not containing calcium. It will also evaluate the association between δ44/42Ca and established biomarkers of bone formation and repair.

The data collected in CALBAL will not by itself allow doctors to decide whether δ44/42Ca is good biomarker of bone mineralisation. However, it will provide additional biological and clinical information that will further clarify its usefulness as biomarker for further research. Together with information from previous studies done by the Chief Investigator which measured the typical δ44/42Ca of healthy children and children with CKD and on dialysis, the data collected in CAL-BAL may inform the design of a future randomised trial of standard-of-care compared to an approach where δ44/42Ca results are used to prescribe the amount of medicine containing calcium children with CKD or on dialysis are given.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-17 years
2. Must be in stable Chronic Kidney Disease (CKD) stage 3b-5 (as per the Kidney Disease Improving Global Outcomes classification) or on dialysis for at least 1 month
3. Hyperphosphataemia defined as a serum P above the age-specific normal level as per the Kidney Disease Outcomes Quality Initiative (KDOQI) guideline, or high or normal P levels in a patient already on a P-binder in the preceding 4 weeks
4. On a stable Ca and P diet as assessed by a dietitian and willing to avoid intentional changes in their dairy intake during the trial period
5. Able to give fully informed consent/ assent as applicable.

Exclusion Criteria:

1. Pre-existing inherited bone disease
2. Glucocorticoid therapy in the preceding year, or a lifetime cumulative steroid exposure ≥6 months
3. Bisphosphonate therapy at any time in the past
4. On cinacalcet in the preceding 6-months
5. Any acute illness in the preceding 2 weeks (when the child was unable to maintain their usual diet or had bed-rest)
6. Living-donor renal transplant planned ≤6 months
7. At screening the albumin-corrected serum calcium cannot be <2.0mMol/L or >2.8mMol/L
8. Already participating in any interventional clinical trial or last trial completed less than 4 weeks previously
9. Previously documented poor compliance with medications
10. Any other contraindication to usual prescription of calcium carbonate or sevelamer carbonate
11. Any other reason in the opinion of the Investigator that the participant may not be suitable
12. Estimated GFR (eGFR) more than 45ml/min/1.73m2
13. Pregnant or lactating
14. Currently on sevelamer (includes sevelamer carbonate or sevelamer hydrochloride)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Ca isotope ratios in serum measured by dual-tracer stable isotope method (Ca isotope fractions δ44/42Ca) of a child after up to 12 weeks treatment with each of two P-binders (Ca based and Ca free). | Measured over 12 weeks. N.B. Treatment changes from sevelamer carbonate to calcium carbonate after 16 weeks in the trial or earlier at the clinician's discretion based on serial monitoring of serum Ca levels.
  Ca isotope ratios in serum measured by dual-tracer stable isotope method (Ca isotope fractions δ44/42Ca) of a child after up to 12 weeks treatment with each of two P-binders (Ca based and Ca free).

SECONDARY OUTCOMES:
Ca isotope ratios in urine measured by dual-tracer stable Ca isotope method (Ca isotope fractions δ44/42Ca) of a child after up to 12 weeks treatment with each of two P-binders (Ca based and Ca free). | Measured over 12 weeks. N.B. Treatment changes from sevelamer carbonate to calcium carbonate after 16 weeks in the trial or earlier at the clinician's discretion based on serial monitoring of serum Ca levels.
  To evaluate the association between the change in δ44/42Ca in blood and urine during treatment with each P-binder with the following quantities (which will also be measured longitudinally):1. Dietary Ca and vitamin D intake (including Ca intake from phosphate binders) 2. Serum Ca, P, PTH, 25(OH)D and 1,25(OH)2D 3. Biomarkers of osteoblast (bone-specific alkaline phosphatase, P1NP), osteoclast (TRAP5b, carboxyterminal cross - linked telopeptide of type I collagen- CTX and NTX), and osteocyte activity (FGF23, sclerostin). 4.To determine the earliest detectable changes in Ca isotope ratios after changing therapy. In children on haemodialysis the Ca isotope ratios will be measured by dual-tracer stable Ca isotope method (Ca isotope fractions δ44/42Ca) in serum and urine (if available) at day 3, day 5, day 8 and day 10 (+/- 2 days) after starting sevelamer carbonate or calcium carbonate.

CONTACTS AND LOCATIONS:
Overall Officials: Rukshana Shroff, MD FRCPCH PhD, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No